CLINICAL TRIAL: NCT02923050
Title: Simple Suppers Scale-up (S3): an Expanded Pilot Study to Determine the Effectiveness of a Family Meals Intervention Aimed at Eliciting Positive Changes in Child Diet and Weight Status
Brief Title: Simple Suppers Scale-up (S3)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Cardinal Health (Industry)
Responsible Party: Principal Investigator, Carolyn Gunther, Assistant Professor, Ohio State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2014B0494
Record Dates: First submitted 2016-09-28; First posted 2016-10-04 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Waitlist control (No Intervention)
- 10-week family meals program (Experimental)
  Interventions: Behavioral: Simple Suppers

INTERVENTIONS:
Behavioral: Simple Suppers — Theory-based 10-week family meals program
  Arms: 10-week family meals program

SUMMARY:
The purpose of this study is to determine effectiveness of a family meals intervention, Simple Suppers, aimed at eliciting positive changes in child dietary intake and weight status.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers: Primary food preparer in the home; responsible for at least one child 4-10 years of age; speak English as the primary language in the home; lived in the U.S. for at least one year.

Exclusion Criteria:

* Family member: Following a restrictive or therapeutic diet.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 223 (Actual)
Dates: Start 2015-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Child standardized body mass index (BMI) | Change from baseline child BMI at 10 weeks

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gunther C, Rogers C, Holloman C, Hopkins LC, Anderson SE, Miller CK, Copeland KA, Dollahite JS, Pratt KJ, Webster A, Labyk AN, Penicka C. Child diet and health outcomes of the simple suppers program: a 10-week, 2-group quasi-experimental family meals trial. BMC Public Health. 2019 Dec 10;19(1):1657. doi: 10.1186/s12889-019-7930-7. PMID 31823753
- [Derived] Rogers C, Anderson SE, Dollahite JS, Hill TF, Holloman C, Miller CK, Pratt KJ, Gunther C. Methods and design of a 10-week multi-component family meals intervention: a two group quasi-experimental effectiveness trial. BMC Public Health. 2017 Jan 9;17(1):50. doi: 10.1186/s12889-016-3908-x. PMID 28069006